CLINICAL TRIAL: NCT04214834
Title: Pragmatic, Randomized, Blinded Trial to Shorten Pharmacologic Treatment of Newborns With Neonatal Opioid Withdrawal Syndrome (NOWS)
Brief Title: Trial to Shorten Pharmacologic Treatment of Newborns With Neonatal Opioid Withdrawal Syndrome (NOWS)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Trials in Neonatal Opioid Withdrawal (ACT NOW) Program (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACTNOW-02
Record Dates: First submitted 2019-12-05; First posted 2020-01-02 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-01

CONDITIONS: Neonatal Opioid Withdrawal Syndrome
Keywords: NOWS
MeSH Terms: interventions — Morphine; Methadone

STUDY DESIGN:
Intervention Model Description: The study will have two intervention arms (rapid-wean and slow-wean) with 251 morphine/methadone treated infants per intervention arm, for a total of 502 morphine/methadone treated infants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy will track dose levels to know where an infant is within a rapid- or slow-wean intervention arm. The clinical team will be blinded to the dose level and will only be aware of the study steps. Both the rapid- and slow-wean intervention arms are depicted to indicate that if each intervention arm has the same number of escalations, the study steps will be identical. This is critical to maintaining the clinical team blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid-wean (Active Comparator): 15% decrements from the stabilization dose of morphine/methadone
  Interventions: Drug: Morphine; Drug: Methadone
- Slow-wean (Active Comparator): 10% decrements from the stabilization dose of morphine/methadone
  Interventions: Drug: Morphine; Drug: Methadone

INTERVENTIONS:
Drug: Morphine — The dose interval for morphine will be either every 3 or 4 hours, per hospital practice. Clinical teams are asked to wean study drug at least every 24 hours.
Drug: Methadone — The dose interval for methadone will be every 8 or 12 hours, per hospital practice. Clinical teams are asked to wean study drug at least every 24 hours.

SUMMARY:
The objective of this study is to evaluate the efficacy of a rapid wean intervention compared with a slow-wean intervention in reducing the number of days of opioid treatment from the first dose of weaning to cessation of opioid among infants receiving an opioid (defined as morphine or methadone) as the primary treatment for neonatal opioid withdrawal syndrome (NOWS).

DETAILED DESCRIPTION:
This will be a pragmatic, randomized, blinded trial comparing a rapid-wean intervention (15% decrements from the stabilization dose) to a slow-wean intervention (10% decrements from the stabilization dose) to determine whether rapid weaning will reduce the number of treatment days among infants receiving morphine or methadone orally as the primary treatment for NOWS. Participating hospitals must provide pharmacologic treatment to at least an average of 12 opioid exposed infants each year, use a scoring system to assess for signs of NOWS (original or modified Finnegan Neonatal Abstinence Scoring system, Eat-Sleep or Console), and provide opioid replacement therapy with either morphine or methadone as the primary drug for treating NOWS. Hospitals may change use of these two opioids during the trial period. The investigators will stratify randomization by hospital.

The study protocol will commence after NOWS signs have been controlled with an opioid (stabilization) and weaning of pharmacologic treatment is to be started. At or before each 24-hour interval, clinical team members will evaluate and score infants, per hospital practice, for signs of NOWS to determine if the infant will tolerate weaning of the study drug. After study drug cessation, the clinical team will observe infants in the hospital for at least 48 hours prior to discharge, which is similar to clinical practice. A trained examiner will administer the Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale (NNNS) to assess neurobehavioral profiles after infants cease study drug and prior to discharge.

At one month post discharge, primary caregivers will complete the Brief Symptom Inventory (BSI), the Maternal Postnatal Attachment Questionnaire (MPAQ) and a caregiver questionnaire. The site research team will contact the primary caregiver(s) to update contact information and/or complete questionnaires when the infant is 6 months, 12 months, 18 months, and 24 months of age. The questionnaires will assess infant wellness, neurobehavioral functioning and development, postnatal attachment and bonding, and caregiver well-being. At 24 months, the infants will be seen during which a, certified developmental specialists, blinded to the intervention, will administer the Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-4) to assess infant neurodevelopment. The BSI and the Brief Infant Toddler Social Emotional Assessment (BITSEA) will also be administered during the 24 month visit along with measures of growth.

ELIGIBILITY:
Inclusion Criteria:

* Hospital Level

  1. Hospital provides pharmacologic treatment to at least an average of 12 opioid exposed infants each year
  2. Hospital uses a scoring system to assess for signs of NOWS (original or modified Finnegan Neonatal Abstinence Scoring system, Eat-Sleep or Console)
  3. Hospital provides opioid replacement therapy with either morphine or methadone as part of pharmacologic treatment of NOWS
* Infant Level

  1. Gestational age ≥ 36 weeks
  2. Receiving scheduled pharmacological therapy with morphine or methadone as the primary drug treatment for NOWS secondary to maternal opioid use
  3. Tolerating enteral feeds and medications by mouth

Exclusion Criteria:

* Hospital Level

  1. Hospitals discharge > 10% of infants from the hospital on opioid replacement therapy on average per year
* Infant Level

  1. Major birth defect (e.g. gastroschisis)
  2. Any major surgery (minor surgery [e.g., circumcision, digit ligation, frenulectomy] is not an exclusion criterion)
  3. Hypoxic-ischemic encephalopathy
  4. Seizures from etiologies other than NOWS
  5. Treatment with opioids for reasons other than NOWS
  6. Respiratory support (nasal cannula or greater) for > 72 hours
  7. Planned discharge from the hospital on opioids
  8. Use of other opioids (e.g., buprenorphine) as primary drugs for treatment of NOWS
  9. Weaning of morphine or methadone as the primary treatment of NOWS has started

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Abhik Das, PhD, Principal Investigator — RTI International; Abbot Laptook, MD, Principal Investigator — Women and Infants Hospital of Rhode Island; Adam Czynski, DO, Principal Investigator — Connecticut Children's Medical Center
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - University of Iowa, Iowa City, Iowa
  - Ochsner Medical Regional Hospital, Kenner, Louisiana
  - Tulane University Health Science Center, New Orleans, Louisiana
  - Ochsner Baptist Clinical Trials Unit, New Orleans, Louisiana
  - MedStar Franklin Square, Hyattsville, Maryland
  - University of Massachusetts Memorial Medical Center-West Campus, Worcester, Massachusetts
  - Central Michigan University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - RTI International, Durham, North Carolina
  - Metrohealth, Cleveland, Ohio
  - Nationwide Childeren's Hospital, Columbus, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Sanford Health, Sioux Falls, South Dakota
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available in NICHD Data and Specimen Hub (DASH).
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Czynski A, Laptook A, Das A, Smith B, Simon A, Greenberg R, Annett R, Lee J, Snowden J, Pedroza C, Lester B, Eggleston B, Bremer D, McGowan E. Pragmatic, randomized, blinded trial to shorten pharmacologic treatment of newborns with neonatal opioid withdrawal syndrome (NOWS). Trials. 2023 Jul 21;24(1):466. doi: 10.1186/s13063-023-07378-x. PMID 37480087

RESULTS

PARTICIPANT FLOW:
Groups:
- Rapid Wean: Rapid Wean: 15% decrements from the stabilization dose of morphine/methadone
- Slow Wean: Slow Wean: 10% decrements from the stabilization dose of morphine/methadone
Period: Overall Study
Arm/Group | Rapid Wean | Slow Wean
Started | 98 | 91
Completed (Completed Intervention) | 94 | 91
Not Completed | 4 | 0
Not completed — Withdrawal by Parent(s)/Legal Guardian(s) | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapid Wean | Slow Wean | Total
Number analyzed (Participants) | 98 | 91 | 189
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 38.8 (1.2) | 38.8 (1.3) | 38.8 (1.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 58 | 56 | 114
  Missing | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or AlaskaNative | 3 | 1 | 4
  Black or African American | 16 | 10 | 26
  Missing | 1 | 1 | 2
  More than one race | 0 | 1 | 1
  Unknown | 4 | 4 | 8
  White | 74 | 74 | 148
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 18 | 35
  Missing | 1 | 1 | 2
  Not Hispanic or Latino | 77 | 66 | 143
  Unknown | 3 | 6 | 9
Mothers opioid treatment [Count of Participants; unit: Participants]
  Buprenorphine w/wo naloxone | 40 | 30 | 70
  Methadone | 32 | 38 | 70
  Missing | 1 | 1 | 2
  None/Other | 25 | 22 | 47
Stabilization dose: Morphine [Mean (Inter-Quartile Range); unit: mg] | 0.22 [0.15 to 0.29] | 0.25 [0.16 to 0.32] | 0.23 [0.15 to 0.30]
Stabilization dose: Methadone [Mean (Inter-Quartile Range); unit: mg] | 0.28 [0.19 to 0.36] | 0.33 [0.20 to 0.38] | 0.31 [0.19 to 0.37]
Infant feed [Count of Participants; unit: Participants]
  unknown | 7 | 3 | 10
  Bottle | 76 | 80 | 156
  Breast | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Days of Opioid Treatment From First Wean to Cessation
Description: The number of days of opioid treatment (used as primary treatment), including escalation, resumption, and spot treatment, from the first weaning dose to cessation of opioid. From the start of opioid study medication until weaning. Infants will exit the study intervention without unblinding (remain in the trial) if they have not weaned off study drug by 35 days (inclusive of the 35th day) form the first weaning dose. Outcome will be truncated at 35 days regardless of the study arm.We note that primary outcome data is missing for 4 participants resulting in total sample of 185 for the primary analysis.
Time Frame: From the start of opioid study medication until weaning. Infants exited the study intervention without unblinding (remained in the trial) by 35 days from the first weaning dose. Outcome truncated at 35 days regardless of the study arm.
Population: An intent-to-treat (ITT) analysis which included all infants participants who were randomized and who provided outcome data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rapid Wean | Slow Wean
Number analyzed (Participants) | 94 | 91
days | 9.3 (6.3) | 11.7 (6.1)
Statistical Analysis 1: Comparison: Rapid Wean vs Slow Wean; A logarithmic transformation was applied to the outcome, centers were added as random effects to account for variation between them; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 2.96, 95% CI 2-sided [1.70 to 4.29] — Given that the model was on the log scale, mean difference and 95% confidence interval were derived from 1,000 bootstrap resamples

2. Secondary Outcome: Days of Opioid Treatment From First Wean to Cessation Among Infants That Were Not Withdrawn in High Enrolling Centers
Description: The number of days of opioid treatment from first wean to cessation among infants that were not withdrawn in high enrolling centers
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rapid Wean | Slow Wean
Number analyzed (Participants) | 65 | 69
days | 8.1 (4.9) | 10.5 (4.2)

3. Secondary Outcome: Days of Opioid Treatment From First Wean to Cessation Among High Enrolling Centers
Description: The number of days of opioid treatment from first wean to cessation among high enrolling centers
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rapid Wean | Slow Wean
Number analyzed (Participants) | 72 | 76
days | 9 (5.9) | 11.3 (5.7)

4. Secondary Outcome: Days of Opioid Treatment From First Wean to Cessation Among Infants That Were Not Withdrawn
Description: The number of days of opioid treatment from first wean to cessation among infants that were not withdrawn
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rapid Wean | Slow Wean
Number analyzed (Participants) | 80 | 79
days | 8 (4.8) | 10.7 (4.1)

ADVERSE EVENTS:
Time Frame: Randomization through 8-weeks post discharge
Arm/Group | Rapid Wean | Slow Wean
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/91
Serious Adverse Events (participants affected / at risk) | 1/98 | 1/91
Other Adverse Events (participants affected / at risk) | 3/98 | 4/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Wean (N=98) | Slow Wean (N=91)
Epidural hematoma (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Skull fracture (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapid Wean (N=98) | Slow Wean (N=91)
Inguinal hernia/repair (Gastrointestinal disorders) | 0 (0) | 1 (1)
Over-sedation (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory disturbances (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Study Protocol (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT04214834/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT04214834/SAP_001.pdf
  • Informed Consent Form: ICF Template (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04214834/ICF_002.pdf
  • Informed Consent Form: Parental Informed Consent and Assent (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04214834/ICF_003.pdf
  • Informed Consent Form: Caregiver-only Consent (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT04214834/ICF_004.pdf
  • Informed Consent Form: Infant-only Consent (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT04214834/ICF_005.pdf